CLINICAL TRIAL: NCT00374842
Title: A Study to Evaluate the Immunogenicity, Safety and Reactogenicity of Adjuvanted Influenza Vaccine Candidates Compared to Fluarix™ Administered Intramuscularly in Subjects Aged 18-59 Years.
Brief Title: Study to Evaluate the Immunogenicity and Safety of 2 Formulations of GlaxoSmithKline (GSK) Biologicals' GSK1247446A Low Dose Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 108656
Record Dates: First submitted 2006-09-08; First posted 2006-09-12 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza vaccine; Prophylaxis Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- GSK1247446A Formulation 1 Group (Experimental): Subjects aged 18 - 59 years at the time of enrolment received one dose of the GSK1247446A vaccine adjuvanted with a full dose of adjuvant at Day 0. The adjuvanted GSK1247446A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK1247446A
- GSK1247446A Formulation 2 Group (Experimental): Subjects aged 18 - 59 years at the time of enrolment received one dose of the GSK1247446A vaccine adjuvanted with a half dose of adjuvant at Day 0. The adjuvanted GSK1247446A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK1247446A
- Fluarix Group (Active Comparator): Subjects aged 18 - 59 years at the time of enrolment received one dose of the Fluarix™ vaccine at Day 0. The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Fluarix™ — GlaxoSmithKline Biologicals' licensed influenza vaccine
  Arms: Fluarix Group
Biological: GSK1247446A — Low-dose GlaxoSmithKline Biologicals' GSK1247446A influenza vaccine
  Arms: GSK1247446A Formulation 1 Group; GSK1247446A Formulation 2 Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of candidate vaccines compared to Fluarix™ administered intramuscularly in subjects aged 18-59 years

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18-59 years at the time of the first vaccination.
* Free of obvious health problems

Exclusion Criteria:

* Use of non-registered products
* Administration of immune-modifying drugs.
* Administration of vaccine 30 days before enrolment in study.
* Immunosuppressive or immunodeficient condition.
* Hypersensitivity to a previous dose of influenza vaccine
* Previous vaccination against influenza in 2006
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* History of confirmed influenza infection within the last 12 Months.
* Acute disease at the time of enrolment/vaccination.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-10-03; Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 108656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 subjects were enrolled in the study. Study duration was of approximately 1 month (30 days) for all subjects.
Period: Overall Study
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Started | 100 | 100 | 100
Completed | 100 | 100 | 100
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (13.94) | 35.0 (13.26) | 37.7 (13.75) | 36.7 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 60 | 57 | 182
  Male | 35 | 40 | 43 | 118

OUTCOME MEASURES:

1. Primary Outcome: Titers of Serum Haemagglutination-inhibition (HI) Antibodies Against Each of the 3 Influenza Strains Assessed.
Description: Influenza strains assessed were the A/New Caledonia (A/CAL), A/Wisconsin (A/WIS), B/Malaysia (B/MAL) strains. Titers were presented as geometric mean titers (GMTs) calculated on subjects with available results, and expressed in haemagglutination-inhibition unit (HIU), e. g. the dilution of a serum haemagglutination-inhibition containing the specific antibody each of the assessed influenza strains at which the solution retained the minimum level of activity needed to neutralize or precipitate the corresponding influenzae antigen. The seropositivity cut-off value of the assay was 10 HIU.
Time Frame: At Day 0 and at Day 21.
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: HIU
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 99 | 99 | 98
HIU
  A/CAL, Day 0 | 31.9 [23.5 to 43.4] | 36.1 [26.9 to 48.5] | 26.1 [20.5 to 33.2]
  A/CAL, Day 21 | 475.4 [352.2 to 641.6] | 399.0 [294.7 to 540.2] | 380.6 [274.2 to 528.4]
  A/WIS, Day 0 | 16.8 [13.1 to 21.5] | 19.9 [15.2 to 25.9] | 14.7 [11.6 to 18.6]
  A/WIS, Day 21 | 276.2 [223.5 to 341.3] | 241.9 [192.9 to 303.4] | 172.3 [136.4 to 217.6]
  B/MAL, Day 0 | 20.4 [15.9 to 26.1] | 22.2 [17.6 to 27.9] | 26.5 [20.9 to 33.6]
  B/MAL, Day 21 | 268.6 [221.3 to 326.0] | 301.5 [246.1 to 369.4] | 219.2 [171.4 to 280.2]

2. Primary Outcome: Number of Seroprotected Subjects Against Each of the 3 Influenza Strains Assessed.
Description: A seroprotected subject was a subject whose antibody titer against each of the influenza strains assessed (A/New Caledonia (A/CAL), A/Wisconsin (A/WIS) and B/Malaysia (B/MAL) strains) was equal to or higher than (>=) the assay seroprotection cut-off value of 40 haemagglutination-inhibition units (HIU) (e. g. the dilution of a serum haemagglutination-inhibition containing the specific antibody each of the assessed influenza strains at which the solution retained the minimum level of activity needed to neutralize or precipitate the corresponding influenzae antigen).
Time Frame: At Day 0 and at Day 21.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 99 | 99 | 98
Subject
  A/CAL, Day 0 | 41 | 55 | 35
  A/CAL, Day 21 | 95 | 97 | 93
  A/WIS, Day 0 | 32 | 37 | 25
  A/WIS, Day 21 | 97 | 97 | 93
  B/MAL, Day 0 | 31 | 39 | 44
  B/MAL, Day 21 | 97 | 98 | 94

3. Primary Outcome: Number of Seroconverted Subjects Against Each of the 3 Influenza Strains Assessed
Description: Influenza strains assessed were the A/New Caledonia (A/CAL), A/Wisconsin (A/WIS), and B/Malaysia (B/MAL) strains. A seroconverted subject was a subject who had either a pre-vaccination serum HI antibody titer lower than 10 haemagglutination-inhibition units (HIU) (e. g. the dilution of a serum haemagglutination-inhibition containing the specific antibody each of the assessed influenza strains at which the solution retained the minimum level of activity needed to neutralize or precipitate the corresponding influenzae antigen) and a post-vaccination titer higher than or equal to 40 HIU, or a pre-vaccination titer >= 10 and at least a four-fold increase in post- vaccination titer.
Time Frame: At Day 21.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 99 | 99 | 98
Subject
  A/CAL, Day 21 | 69 | 64 | 66
  A/WIS, Day 21 | 88 | 79 | 73
  B/MAL, Day 21 | 76 | 82 | 65

4. Primary Outcome: Seroconversion Factor Against Each of the 3 Influenza Strains Assessed.
Description: Influenza strains assessed were the A/New Caledonia (A/CAL), A/Wisconsin (A/WIS), and B/Malaysia (B/MAL) strains. The seroconversion factor (SCF) was defined as a ratio, as the fold increase in serum haemagglutination-inhibition geometric mean titers (GMTs) post-vaccination compared to Day 0 (with GMTs in the above calculation expressed in haemagglutination-inhibition units (HIU) [e. g. the dilution of a serum haemagglutination-inhibition containing the specific antibody each of the assessed influenza strains at which the solution retained the minimum level of activity needed to neutralize or precipitate the corresponding influenza antigen]).
Time Frame: At Day 21.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Groups:
- GSK1247446A Formulation 2 Group: Subjects aged 18 - 59 years at the time of enrolment received one dose of the GSK1247446A vaccine adjuvanted with a full dose of adjuvant at Day 0. The adjuvanted GSK1247446A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 99 | 99 | 98
Fold increase
  A/CAL, Day 21 | 14.9 [10.4 to 21.3] | 11.0 [7.7 to 15.9] | 14.6 [9.9 to 21.6]
  A/WIS, Day 21 | 16.5 [13.0 to 20.9] | 12.2 [9.2 to 16.1] | 11.7 [8.8 to 15.6]
  B/MAL, Day 21 | 13.2 [10.0 to 17.4] | 13.6 [10.2 to 18.0] | 8.3 [6.2 to 11.0]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling the site of injection. Any = occurrence of a solicited local symptom regardless of intensity grade. Grade 3 pain = Pain which prevented normal activity. Grade 3 ecchymosis/redness/swelling = ecchymosis/redness/swelling at injection site with a diameter larger than (>) 50 millimeters (mm). All solicited local symptoms assessed were considered by the investigator as causally related to the study vaccination.
Time Frame: Within the 7-day follow-up period (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 100 | 100 | 100
Subject
  Any ecchymosis | 6 | 11 | 6
  Grade 3 ecchymosis (> 50 mm) | 0 | 0 | 0
  Any pain | 92 | 89 | 64
  Grade 3 pain | 10 | 0 | 0
  Any redness | 24 | 12 | 15
  Grade 3 redness (> 50 mm) | 6 | 2 | 1
  Any swelling | 28 | 17 | 7
  Grade 3 swelling (> 50 mm) | 7 | 4 | 2

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever (axillary temperature higher than or equal to (>=) 37.5 degrees Celsius (°C)), headache, muscle aches, and shivering. Any = Occurrence of a particular symptom regardless of intensity or relationship to vaccination. Grade 3 symptom = Symptom which prevented normal activity. Related = Symptom assessed by the investigator as causally related to the study vaccination. Grade 3 fever = axillary temperature higher than 39.0°C.
Time Frame: Within the 7-day follow-up period (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 100 | 100 | 100
Subject
  Any arthralgia | 32 | 14 | 7
  Grade 3 arthralgia | 3 | 1 | 0
  Related arthralgia | 32 | 13 | 5
  Any fatigue | 60 | 42 | 28
  Grade 3 fatigue | 6 | 2 | 1
  Related fatigue | 59 | 39 | 26
  Axillary fever (>= 37.5°C) | 30 | 12 | 2
  Grade 3 axillary fever (> 39.0°C) | 2 | 0 | 0
  Related axillary fever (>= 37.5°C) | 30 | 12 | 2
  Any headache | 51 | 40 | 29
  Grade 3 headache | 9 | 6 | 3
  Related headache | 50 | 35 | 23
  Any muscle aches | 48 | 30 | 12
  Grade 3 muscle aches | 4 | 2 | 0
  Related muscle aches | 47 | 29 | 11
  Any shivering | 33 | 13 | 5
  Grade 3 shivering | 2 | 2 | 0
  Related shivering | 33 | 13 | 5

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. Any AE = any occurrence of an AE, regardless of intensity or relationship to study vaccination. Grade 3 = an event that prevented normal activity. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within the 30-day follow-up period (Days 0-29) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 100 | 100 | 100
Subject
  Subject(s) with any unsolicited AE(s) | 55 | 47 | 35
  Subject(s) with Grade 3 unsolicited AE(s) | 11 | 5 | 6
  Subject(s) with related unsolicited AE(s) | 33 | 22 | 16

8. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE = any occurrence of an SAE, regardless of relationship to study vaccination. A related SAE = an SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: From study start to study end, from Day 0 to Day 30
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Number analyzed (Participants) | 100 | 100 | 100
Subject
  Subject(s) with any SAE(s) | 1 | 0 | 0
  Subject(s) with related SAE(s) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within the 7-day (Days 0-6) follow-up period after vaccination. Unsolicited adverse events: Within the 30-day (Days 0-29) follow-up period after vaccination. Serious adverse events: From study start to study end (Days 0-30)
Arm/Group | GSK1247446A Formulation 1 Group | GSK1247446A Formulation 2 Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 98/100 | 95/100 | 81/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Formulation 1 Group (N=100) | GSK1247446A Formulation 2 Group (N=100) | Fluarix Group (N=100)
Post procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Formulation 1 Group (N=100) | GSK1247446A Formulation 2 Group (N=100) | Fluarix Group (N=100)
Ecchymosis (General disorders) | 6 | 11 | 6
Pain (General disorders) | 92 | 89 | 64
Redness (General disorders) | 24 | 12 | 15
Swelling (General disorders) | 28 | 17 | 7
Arthralgia (General disorders) | 32 | 14 | 7
Fatigue (General disorders) | 60 | 42 | 28
Headache (General disorders) | 51 | 40 | 29
Muscle aches (General disorders) | 48 | 30 | 12
Shivering (General disorders) | 33 | 13 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 2
Nasopharyngitis (Infections and infestations) | 15 | 8 | 11
Headache (Nervous system disorders) | 9 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.